CLINICAL TRIAL: NCT02681510
Title: UW-CTRI Smoking Cessation Medication Tolerability Study
Brief Title: UW-CTRI Triple Medication Smoking Cessation Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 2015-1376
Record Dates: First submitted 2016-02-09; First posted 2016-02-12 (Estimated); Results first posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-09

CONDITIONS: Smoking
Keywords: medication tolerability
MeSH Terms: conditions — Smoking | interventions — Varenicline; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Three drug intervention (Experimental): varenicline, nicotine patch and nicotine lozenge for 12 weeks
  Interventions: Drug: Varenicline; Drug: Nicotine Transdermal Patch; Drug: Nicotine Mini

INTERVENTIONS:
Drug: Varenicline — Standard FDA approved 12 weeks of treatment with Varenicline
  Other Names: Chantix
Drug: Nicotine Transdermal Patch — Standard FDA approved 12 weeks of treatment with Nicotine Transdermal Patch
Drug: Nicotine Mini — Standard FDA approved 12 weeks of treatment with Nicotine Mini-Lozenge
  Other Names: Nicotine Mini-Lozenge

SUMMARY:
This study will focus on enhancing future smoking cessation treatment effectiveness by piloting a potentially more powerful combination of three FDA-approved pharmacotherapies: varenicline plus combination of two types of nicotine replacement therapy (NRT) treatment (nicotine lozenge and nicotine patch). Data from this pilot study will help inform the design of future studies that would use this combination treatment as a cessation tool within the chronic care arsenal of treatments.

DETAILED DESCRIPTION:
Recent research suggests that a new combination therapy may be especially effective in increasing long-term abstinence from smoking. A key purpose of the proposed study is to examine what types of tolerability concerns, if any, emerge from the simultaneous use of three FDA-approved cessation medications (varenicline, nicotine patch, and nicotine lozenge) and the timing of those events, in order to better assess how the use of this combination of tobacco cessation medicines can be most effectively and safely delivered and monitored. Study participants will take the three medications for 12 weeks in a manner consistent with labeling. Adverse events will be assessed at all study visits.

ELIGIBILITY:
Inclusion Criteria:

* Age >17 years;
* >=5 cigarettes/day for the previous 6 months;
* alveolar CO >= 6 ppm; able to read, write and speak English;
* planning to remain in the intervention catchment area for at least 4 months; not currently taking bupropion or varenicline;
* if the participant is currently using NRT, s/he agrees to use only study medication for the duration of the study;
* free of medical contraindications to NRT and varenicline; and,
* if participant is a woman of childbearing potential, using an approved method of birth control during treatment.

Exclusion Criteria:

* Current diagnosis of/treatment for psychosis or bipolar disorder;
* suicidal ideation within the past 12 months; any history of suicide attempts; * significant hepatic or renal impairment; history of significant allergic reactions to varenicline or any type of NRT in the past;
* use of any investigational drugs in the previous 30 days. -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-06-13 (Actual); Study Completion 2016-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Fiore, Principal Investigator — University of Wisconsin--CTRI
Locations (1):
- UW CTRI, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Berg KM, Jorenby DE, Baker TB, Fiore MC. Triple Smoking Cessation Therapy with Varenicline, Nicotine Patch and Nicotine Lozenge: A Pilot Study to Assess Tolerability, Satisfaction, and End-of-Treatment Quit Rates. J Smok Cessat. 2018 Sep;13(3):145-153. doi: 10.1017/jsc.2017.18. Epub 2017 Sep 25. PMID 30524509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via Facebook ads contextually tagged to appear only to adults in the Madison, WI area who had "liked" or posted about smoking.
Period: Overall Study
Arm/Group | Three Drug Intervention
Started | 36
Completed | 26
Not Completed | 10
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Arm/Group | Three Drug Intervention
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33
  African-American | 1
  Asian | 1
  Unknown | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Assess adverse event rates in relation to participant ability to continue use of all 3 medications throughout the treatment period
Time Frame: 12 weeks
Population: All study participants (N=36)
Measure: Count of Participants; unit: Participants
Arm/Group | Three Drug Intervention
Number analyzed (Participants) | 36
Participants
  Insomnia | 27
  Vivid Dreams | 26
  Nausea | 23
  Mood Changes | 15
  Dizziness | 14
  Skin Rash | 7
  Sweating | 7
  Shortness of Breath | 5
  Vomiting | 5
  Chest Tightness | 4
  Angina | 1

2. Secondary Outcome: Participant Satisfaction With Medications' Ability to Control Withdrawal Symptoms
Description: Satisfaction with Medications' Ability to Control Withdrawal Symptoms assessed on a 1-10 Likert Scale (higher value=greater satisfaction)
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Three Drug Intervention
Number analyzed (Participants) | 36
units on a scale | 9.1 (1.2)

3. Secondary Outcome: Participant Satisfaction With Medications' Ability to Help Participant Quit Smoking
Description: Participant Satisfaction with Medications' Ability to Help Participant Quit Smoking assessed on a 1-10 Likert Scale (higher value=greater satisfaction)
Time Frame: Week 12
Population: All study participants (N=36)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Three Drug Intervention
Number analyzed (Participants) | 36
units on a scale | 9.2 (1.4)

4. Secondary Outcome: Number of Participants Who Reported Quitting at the End of Treatment
Description: Self-reported Quit Rate at End of Treatment (12 Weeks); assessed as no smoking in the 7 days prior to the Week 12 follow-up call
Time Frame: Week 12
Population: All study participants (N=36)
Measure: Count of Participants; unit: Participants
Arm/Group | Three Drug Intervention
Number analyzed (Participants) | 36
Participants | 21

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The AE assessment specifically queried the presence or absence of: chest tightness, angina, dizziness, dreams, insomnia, mood changes, nausea, skin rash, sweating, shortness of breath, and vomiting. The severity of each AE was graded as: mild (no interference with daily activities, no medications needed to treat symptom); moderate (some interference with daily activities, over-the-counter medications needed); severe (unable to perform daily activity, prescription medication needed).
Arm/Group | Three Drug Intervention
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 35/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Three Drug Intervention (N=36)
Insomnia (Psychiatric disorders) | 27 (27)
Vivid Dreams (Psychiatric disorders) | 26 (26)
Nausea (Gastrointestinal disorders) | 23 (23)
Mood Changes (Psychiatric disorders) | 15 (15)
Dizziness (Nervous system disorders) | 14 (14)
Skin Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Sweating (General disorders) | 7 (7)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 5 (5)
Chest Tightness (Cardiac disorders) | 4 (4)
Angina (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-01-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT02681510/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-01-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT02681510/Prot_SAP_001.pdf